CLINICAL TRIAL: NCT05442996
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of HLX35 (Recombinant Humanized Anti-EGFR and Anti-4-1BB Bispecific Antibody Injection) in Combination With HLX10 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of HLX35 in Combination With HLX10 in Patients With Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLX35HLX10-101
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX35+HLX10 (Experimental): Subjects will receive HLX35 in combination with HLX10 therapy, every 2 weeks as one treatment cycle.
  Interventions: Drug: HLX35; Drug: HLX10

INTERVENTIONS:
Drug: HLX35 — The dose of HLX35 is set at 0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg, and 10 mg/kg. It is administered intravenously every 2 weeks on day 1 of each cycle.
  Other Names: Recombinant humanized anti-EGFR and anti-4-1BB bispecific antibody injection
Drug: HLX10 — The dose of HLX10 is fixed at 200 mg. It is administered intravenously once every 2 weeks on day 1 of each cycle.
  Other Names: Recombinant humanized anti-PD-1 monoclonal antibody injection

SUMMARY:
This is a phase I clinical study designed to evaluate the safety, tolerability, PK characteristics, and preliminary efficacy of HLX35 in combination with HLX10 in patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
For HLX35, 5 dose levels are set, starting at 0.1 mg/kg, q2w, followed by gradually escalating doses of 0.3 mg/kg, 1 mg/kg, 3 mg/kg, and 10 mg/kg; for HLX10, a fixed dose of 200 mg is set, q2w, without dose escalation. The "3 + 3" design is used for dose escalation in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the clinical study; be able to sign the ICF based on full understanding and awareness of the study; have the willingness to follow and the capacity to complete all trial procedures;
2. Aged ≥ 18 years at the time of signing the ICF;
3. Advanced or metastatic solid malignancies confirmed cytologically or histopathologically, prior failure of standard therapy, free of standard therapy or intolerant of standard therapy;
4. Interval between completion of prior systemic anti-tumor treatment (chemotherapy, targeted therapy, and immunotherapy) and the first dose in this study is ≥ 28 days; interval between completion of endocrine or TCM anti-tumor therapy and the first dose in this study is ≥ 14 days; interval between completion of any other anti-tumor treatment with clinical study drug and the first dose in this study is ≥ 28 days;
5. Prior anti-tumor treatment-related AE recovering to grade ≤ 1 as per CTCAE v5.0 prior to the first dose (except for alopecia);
6. At least one measurable target lesion assessed by the investigator according to the RECIST v1.1 is required within 4 weeks prior to the first dose (Note: Measurable target lesions may not be selected from the previously irradiated site. If a target lesion at a previously irradiated site is the only optional target lesion, the imaging data before and after significant progression of this lesion after radiotherapy completion should be provided);
7. ECOG performance status score is 0 or 1 within 7 days prior to the first dose;
8. Life expectancy of the patient prior to the first dose judged by the investigator is ≥ 12 weeks;
9. Major organ functions are normal;
10. Women of childbearing potential must complete a serum pregnancy test and have a negative result within 7 days prior to the first dose;
11. Female subjects of childbearing potential or male subjects whose partners are women of childbearing potential must agree to take at least one medically accepted contraceptive measure (intra-uterine device, contraceptive, condom, etc.) from the time of signing the ICF until 6 months after the last dose of the investigational product.

Exclusion Criteria:

1. Other active malignancies within 2 years prior to the first dose of investigational product. Localized tumors that have been cured, such as basal cell carcinoma, squamous-cell skin cancer, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, breast cancer in situ, etc., are acceptable;
2. Patients who are going to receive or have received an organ or bone marrow transplant;
3. Patients with uncontrolled pleural effusion, pericardial effusion, or ascites requiring frequent drainage (monthly or more frequently);
4. Symptomatic brain or meningeal metastases (unless the patient has been treated for > 3 months, there is no evidence of progression on imaging within 4 weeks prior to the first dose, and the tumor-related clinical symptoms are stable);
5. Patients with cerebrovascular accident, myocardial infarction, unstable angina, poorly controlled arrhythmia (including QTc intervals ≥ 450 ms in males and ≥ 470 ms in females) (QTc intervals are calculated by Fridericia formula) occurring within half a year;
6. A cardiac insufficiency of Grade III or IV according to the New York Heart Association (NYHA) classification (Appendix 6), or a left ventricular ejection fraction (LVEF) < 50% based on echocardiography;
7. Human immunodeficiency virus (HIV) infection;
8. Positive (+) for hepatitis B surface antigen (HBsAg) or positive (+) for hepatitis B core antibody (HBcAb), with the hepatitis B virus deoxyribonucleic acid (HBV-DNA) ≥2000 copies /ml, or the presence of active hepatitis determined clinically; hepatitis C (positive for HCV antibody and positive for HCV-RNA);
9. Patients with grade 3-4 drug-related hepatitis;
10. Patients with active pulmonary tuberculosis;
11. Patients with prior and current interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired lung function, etc. that may interfere with the detection and management of suspected drug-related pulmonary toxicity;
12. Patients with known active or suspected autoimmune diseases. Patients who are allowed to have a history of autoimmune disease at enrollment but with no requirement for systemic immunosuppressive therapy at least 12 months prior to screening;
13. Have received treatment with live vaccines within 28 days prior to the first dose. Patients may receive inactivated viral vaccines for seasonal influenza and 2019-nCoV vaccines, but may not receive live attenuated influenza vaccines via intranasal route;
14. Patients requiring treatment with systemic glucocorticoids (> 10 mg/day prednisone efficacy dose) or other immunosuppressive drugs within 14 days prior to the first dose or during the study. However, patients are allowed to be enrolled under the following conditions: in the absence of active autoimmune disease, patients are allowed to use topical or inhaled glucocorticoids and adrenal glucocorticoids replacement therapy at an effective dose equivalent to ≤ 10 mg/day of prednisone;
15. With any serious infection requiring systemic anti-infective therapy within 14 days prior to the first dose of the investigational product;
16. Major surgery within 28 days prior to the first dose of investigational product. A major surgery is defined as a surgery that takes at least 3 weeks of postoperative recovery before receiving treatment in this study;
17. Prior treatment with antibody drugs against immune checkpoint inhibitors (such as PD-1, PD-L1, and CTLA4) or anti-4-1BB antibody drugs;
18. With a history of severe allergy to any monoclonal antibody or any excipient of the investigational product;
19. Pregnant or lactating women;
20. Known history of psychotropic substance abuse or drug use;
21. Have other conditions not suitable for inclusion as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-06 (Estimated); Primary Completion 2024-04-22 (Estimated); Study Completion 2025-04-22 (Estimated)

PRIMARY OUTCOMES:
Number of occurrences and incidence of each adverse event (AE) | up to 2 years
The proportion of patients experiencing dose limiting toxicity (DLT) events | from first dose to the end of Cycle 2 (each cycle is 14 days)
The maximum tolerated dose (MTD) | from first dose to the end of Cycle 2 (each cycle is 14 days)

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | up to 2 years
Time to peak (Tmax) | up to 2 years
Area under the concentration-time curve (AUC) | up to 2 years
Elimination half-life (t1/2) | up to 2 years
Clearance (CL) | up to 2 years
Volume of distribution (Vz) | up to 2 years
Accumulation Index (Rac) | up to 2 years
4-1BB receptor occupancy of T-cells | up to 2 years
soluble 4-1BB level | up to 2 years
incidence of anti-HLX35 antibody (ADA) and its neutralizing antibody (NAb) | up to 2 years
Objective response rate (ORR) | up to 2 years
Disease control rate (DCR) | up to 2 years
Duration of response (DOR) | up to 2 years
Progression-free survival (PFS) | up to 2 years
Overall Survival (OS) | up to 2 years